CLINICAL TRIAL: NCT00280891
Title: Review of Palliative Radiotherapy in the Management of Advanced Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Other Study IDs: 18882
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2006-07

CONDITIONS: Head and Neck Cancer
Keywords: head and neck; cancer; palliation; radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To describe the charactersitics of patients with advanced head and neck cancer treated with palliative intent and determine outcome in terms of symptom control and toxicity

ELIGIBILITY:
Inclusion Criteria:

* squamous cell carcinoma of the head and neck, primary treatment given with palliative intent

Exclusion Criteria:

* radical treatment, palliative treatment following local recurrence, adenocarcinoma, salivary gland carcinoma or melanoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-01; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold Lau, MD, Principal Investigator — Alberta Cancerboard
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada